CLINICAL TRIAL: NCT06762912
Title: The Short-term Effect of Low-load Resistance Training with Blood-flow Restriction on Somatosensory-evoked Potentials in Healthy Young Adults - a Randomized Crossover Trial
Brief Title: The Short-term Effect of Low-load Resistance Training with Blood-flow Restriction on Somatosensory-evoked Potentials in Healthy Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Taif A. M. Omran, Master's Student, University of Sharjah
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: BFRT-SSEP
Record Dates: First submitted 2024-12-23; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: The Current Study Focuses on Investigating the Short-term Effect of BFRT on the Somatosensory System Among Healthy Young Adults
Keywords: Blood Flow Restriction Training; Somatosensory Evoked Potentials; Neuroplasticity; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the three groups: small cuff width (5 cm), medium cuff width (12 cm), and large cuff width (18 cm). Each participant in all three groups will enroll in the three experimental sessions in a random order. All experimental sessions will be provided by the same physiotherapist to minimize the inter-rater variations.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Passive application of BFR cuff (Experimental)
  Interventions: Other: Passive application of BFR cuff
- Resistance exercise with BFR (Experimental)
  Interventions: Other: Resistance exercise with BFR
- Resistance exercise without BFR (Experimental)
  Interventions: Other: Resistance exercise without BFR

INTERVENTIONS:
Other: Passive application of BFR cuff — The first experimental session will start by conducting the one repetition maximum (1-RM) test of unilateral knee extension of the dominant leg, in which the dominant side was identified by asking the participants which side they will use to kick a ball. Before conducting the 1-RM test, 5 minutes warm-up on the cycle ergometer at 75W will be done. Calibration of the dynamometer will be done before operating the machine with each participant, then the participant will be positioned on the dynamometer seat comfortably with ensuring the back is supported and the knee is aligned with the axis of rotation. The participant will be asked to complete one successful repetition of knee extension through full range of motion (ROM), with increasing load until the participant can no longer complete full knee extension ROM, 3 minutes of rest will be allowed between attempts until the 1-RM is identified.
  Arms: Passive application of BFR cuff
Other: Resistance exercise with BFR — For both experimental sessions 2 and 3, the order of exercise condition will be randomly selected, either to be (1) the application of BFR cuff with resistance exercise, or (2) resistance exercise without the application of BFR cuff to decrease the incidence of learning effect. Cuff pressure during the application of BFR will be standardized to 50% of AOP.
  The resistance exercise for both experimental sessions 2 and 3 will be exactly similar and will involve four sets of isometric knee extensions at an intensity of 20% of 1-RM with repetitions of 30, 15, 15, and 15 by using the isokinetic dynamometer machine, which has a good to excellent test-retest reliability for knee extension movement with ICC value of 0.95-0.99. To minimize cognitive and neuromuscular fatigue, the experimental sessions will be separated by a minimum of three days (72 hours).
  Arms: Resistance exercise with BFR
Other: Resistance exercise without BFR — For both experimental sessions 2 and 3, the order of exercise condition will be randomly selected, either to be (1) the application of BFR cuff with resistance exercise, or (2) resistance exercise without the application of BFR cuff to decrease the incidence of learning effect. Cuff pressure during the application of BFR will be standardized to 50% of AOP.
  The resistance exercise for both experimental sessions 2 and 3 will be exactly similar and will involve four sets of isometric knee extensions at an intensity of 20% of 1-RM with repetitions of 30, 15, 15, and 15 by using the isokinetic dynamometer machine, which has a good to excellent test-retest reliability for knee extension movement with ICC value of 0.95-0.99. To minimize cognitive and neuromuscular fatigue, the experimental sessions will be separated by a minimum of three days (72 hours).
  Arms: Resistance exercise without BFR

SUMMARY:
The goal of this clinical trial is to investigate the short-term effect of lower limb BFRT on the somatosensory processing and related changes in SSEP amplitude and latency. The main questions it aims to answer are:

* Is there an effect of short-term application of BFRT on the somatosensory system?
* How do different cuff widths affect the somatosensory system?
* How do three different cuff widths affect perceived pain? Researchers will compare 3 different cuff widths to see if different cuff widths affect the somatosensory system and perceived pain.

Participants will:

* Undergo 3 experimental sessions, sessions will be separated by 72 hours and the order of the sessions to be randomly selected.
* Perform low-load resistance training with blood flow restriction.

DETAILED DESCRIPTION:
The current study will be conducted in the college of health sciences, physiotherapy department, in the medical campus in the University of Sharjah, Sharjah, United Arab Emirates. The study design is a Randomized Crossover Trial, which will include three groups of healthy young adults, each group will use a different cuff widths (small cuff width (5 cm), medium cuff width (12 cm), and large cuff width (18 cm)). Participants in all three groups will undergo three experimental sessions in a random order, which will include the application of a blood flow restriction cuff combined with resistance exercise, the application of a blood flow restriction cuff without resistance exercise, and traditional resistance exercise without a blood flow restriction cuff. During each session, SSEP measurements will be recorded at three time points: before, during, and after the experimental session by stimulating the tibial nerve at the ankle and measuring the SSEP amplitude and latency.

Healthy young adults aged 18-30 years of both genders will be recruited through word of mouth and through social media by sharing the study flyer. Then, they will be screened for their eligibility to participate in the current study. Participants who will meet the eligibility criteria will be asked to provide their consent after the study is explained by filling out the consent form.

Participants will be randomly assigned to one of the three groups: (1) small cuff width (5 cm), (2) medium cuff width (12 cm), and (3) large cuff width (18 cm) by using permuted block randomization method with large, random, and variable block sizes to ensure groups are balanced and selection bias is minimized.

The first experimental session will start by conducting the one repetition maximum (1-RM) test of unilateral knee extension of the dominant leg, in which the dominant side was identified by asking the participants which side they will use to kick a ball. Before conducting the 1-RM test, 5 minutes warm-up on the cycle ergometer at 75W will be done. Calibration of the dynamometer will be done before operating the machine with each participant, then the participant will be positioned on the dynamometer seat comfortably with ensuring the back is supported and the knee is aligned with the axis of rotation. The participant will be asked to complete one successful repetition of knee extension through full range of motion (ROM), with increasing load until the participant can no longer complete full knee extension ROM, 3 minutes of rest will be allowed between attempts until the 1-RM is identified. To eliminate the effect of fatigue after 1-RM test, the first experimental session will always include the application of the BFR cuff without resistance exercise.

For both experimental sessions 2 and 3, the order of exercise condition will be randomly selected, either to be (1) the application of BFR cuff with resistance exercise, or (2) resistance exercise without the application of BFR cuff to decrease the incidence of learning effect. Cuff pressure during the application of BFR will be standardized to 50% of AOP.

The resistance exercise for both experimental sessions 2 and 3 will be exactly similar and will involve four sets of isometric knee extensions at an intensity of 20% of 1-RM with repetitions of 30, 15, 15, and 15 by using the isokinetic dynamometer machine, which has a good to excellent test-retest reliability for knee extension movement with ICC value of 0.95-0.99. To minimize cognitive and neuromuscular fatigue, the experimental sessions will be separated by a minimum of three days (72 hours).

ELIGIBILITY:
Inclusion Criteria:

* Participants will be included if they are aged 18-30 years of both genders, with no history of cardiovascular problems or osteo-articular problems in the lower limbs, and if they responded negatively to all items of the Physical Activity Readiness Questionnaire (PAR-Q).
* Participants will be included if they have a body mass index (BMI) less than 25 or non-overweight individuals.
* Use of the long international physical activity questionnaire (L-IPAQ) to ensure all participants have equal physical activity levels.

Exclusion Criteria:

* Participants will be excluded if they did not meet the inclusion criteria, and if they had a history of deep vein thrombosis (DVT), congenital heart disease, varicose veins, currently pregnant, or any contraindications to exercise.
* Participants will be excluded if they were diagnosed with any neurological disease.
* Participants will be excluded if they have had any musculoskeletal injury in the past 3 months to avoid potential effect on their physical activity levels.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Somatosensory-evoked Potential | 1st Session: Before BFR cuff. During (4 times, 2 min apart). After (4 times, 5 min apart). 2nd & 3rd Sessions: Before exercise with/without BFR cuff. During (4 times, after each set, during rest period). After (4 times, 5 min apart).
  SSEP is a reliable, reproducible, and frequently employed to detect alterations in electrophysiological conduction within the central and peripheral nervous pathways. The assessment of SSEP will involve the placement of electrodes for tibial nerve stimulation at the ankle, which includes both stimulating and recording electrodes.

SECONDARY OUTCOMES:
Perceived Pain | Immediately after each session: - Rate perceived pain during the session (BFR cuff application and resistance exercise). - Rate if they are currently experiencing pain.
  Visual analogue scale (VAS) is widely used to measure the frequency or intensity of various symptoms. VAS is valid, reliable, and frequently used outcome measure to measure intensity of perceived pain. Electronic-based VAS will be used to measure the level of perceived pain after the application of different cuff widths, where there will be a 10-cm/100-mm long horizontal line, with "No pain" to be rated as 0 mm, while "Worst imaginable pain" to be rated as 100 mm and the participant is asked to draw a vertical mark on the horizontal line indicating their level of perceived pain.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sharjah, Sharjah city, United Arab Emirates

REFERENCES:
- [Background] Yusof, N., (2019). Likert Scale vs. Visual analogue scale on vehicle seat discomfort questionnaire: a review. Malaysian Journal of Medicine and Health Sciences, 15(204).
- [Background] Muzyka IM, Estephan B. Somatosensory evoked potentials. Handb Clin Neurol. 2019;160:523-540. doi: 10.1016/B978-0-444-64032-1.00035-7. PMID 31277874
- [Background] Li X, Li J, Qing L, Wang H, Ma H, Huang P. Effect of quadriceps training at different levels of blood flow restriction on quadriceps strength and thickness in the mid-term postoperative period after anterior cruciate ligament reconstruction: a randomized controlled external pilot study. BMC Musculoskelet Disord. 2023 May 8;24(1):360. doi: 10.1186/s12891-023-06483-x. PMID 37158913
- [Background] Wanner M, Probst-Hensch N, Kriemler S, Meier F, Autenrieth C, Martin BW. Validation of the long international physical activity questionnaire: Influence of age and language region. Prev Med Rep. 2016 Mar 9;3:250-6. doi: 10.1016/j.pmedr.2016.03.003. eCollection 2016 Jun. PMID 27419023
- [Background] Korakakis V, Whiteley R, Giakas G. Low load resistance training with blood flow restriction decreases anterior knee pain more than resistance training alone. A pilot randomised controlled trial. Phys Ther Sport. 2018 Nov;34:121-128. doi: 10.1016/j.ptsp.2018.09.007. Epub 2018 Sep 19. PMID 30268966
- [Background] Sousa J, Neto GR, Santos HH, Araujo JP, Silva HG, Cirilo-Sousa MS. Effects of strength training with blood flow restriction on torque, muscle activation and local muscular endurance in healthy subjects. Biol Sport. 2017 Mar;34(1):83-90. doi: 10.5114/biolsport.2017.63738. Epub 2016 Dec 1. PMID 28416903
- [Background] Shousha T, Alayat M, Moustafa I. Effects of low-level laser therapy versus soft occlusive splints on mouth opening and surface electromyography in females with temporomandibular dysfunction: A randomized-controlled study. PLoS One. 2021 Oct 1;16(10):e0258063. doi: 10.1371/journal.pone.0258063. eCollection 2021. PMID 34597318
- [Background] Alghadir AH, Anwer S, Iqbal A, Iqbal ZA. Test-retest reliability, validity, and minimum detectable change of visual analog, numerical rating, and verbal rating scales for measurement of osteoarthritic knee pain. J Pain Res. 2018 Apr 26;11:851-856. doi: 10.2147/JPR.S158847. eCollection 2018. PMID 29731662
- [Background] Cidem M, Sahin Z, Aydin T, Aysal F. Somatosensory evoked potential findings in ankylosing spondylitis. Eurasian J Med. 2014 Feb;46(1):42-6. doi: 10.5152/eajm.2013.100. PMID 25610293
- [Background] Tuominen J, Leppanen M, Jarske H, Pasanen K, Vasankari T, Parkkari J. Test-Retest Reliability of Isokinetic Ankle, Knee and Hip Strength in Physically Active Adults Using Biodex System 4 Pro. Methods Protoc. 2023 Mar 9;6(2):26. doi: 10.3390/mps6020026. PMID 36961046
- [Background] Maudrich T, Degener S, Ragert P, Kenville R. The impact of acute blood-flow-restriction resistance exercise on somatosensory-evoked potentials in healthy adults. Exp Physiol. 2024 Nov;109(11):1869-1881. doi: 10.1113/EP091911. Epub 2024 Sep 4. PMID 39233383
- [Background] Fatela P, Reis JF, Mendonca GV, Avela J, Mil-Homens P. Acute effects of exercise under different levels of blood-flow restriction on muscle activation and fatigue. Eur J Appl Physiol. 2016 May;116(5):985-95. doi: 10.1007/s00421-016-3359-1. Epub 2016 Mar 26. PMID 27017495
- [Background] Ilett MJ, Rantalainen T, Keske MA, May AK, Warmington SA. The Effects of Restriction Pressures on the Acute Responses to Blood Flow Restriction Exercise. Front Physiol. 2019 Aug 13;10:1018. doi: 10.3389/fphys.2019.01018. eCollection 2019. PMID 31456694
- [Background] van Melick N, Meddeler BM, Hoogeboom TJ, Nijhuis-van der Sanden MWG, van Cingel REH. How to determine leg dominance: The agreement between self-reported and observed performance in healthy adults. PLoS One. 2017 Dec 29;12(12):e0189876. doi: 10.1371/journal.pone.0189876. eCollection 2017. PMID 29287067
- [Background] Carter, K., Scheffold, A. L., Renteria, J., Berger, V. W., Luo, Y. A., Chipman, J. J., & Sverdlov, O. (2024). Regulatory Guidance on Randomization and the Use of Randomization Tests in Clinical Trials: A Systematic Review. Statistics in Biopharmaceutical Research, 16(4), 428-440. https://doi.org/10.1080/19466315.2023.2239521
- [Background] Broglio K. Randomization in Clinical Trials: Permuted Blocks and Stratification. JAMA. 2018 Jun 5;319(21):2223-2224. doi: 10.1001/jama.2018.6360. No abstract available. PMID 29872845
- [Background] Patterson SD, Hughes L, Warmington S, Burr J, Scott BR, Owens J, Abe T, Nielsen JL, Libardi CA, Laurentino G, Neto GR, Brandner C, Martin-Hernandez J, Loenneke J. Blood Flow Restriction Exercise: Considerations of Methodology, Application, and Safety. Front Physiol. 2019 May 15;10:533. doi: 10.3389/fphys.2019.00533. eCollection 2019. PMID 31156448